CLINICAL TRIAL: NCT07347613
Title: Long-term Follow-up of Diabetic Patients From the GLUTADIAB Study
Acronym: GlutaDiab2
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A02804-45
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetes
Keywords: glutamine; cardiovascular
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A unique venous blood sampling of 10 tubes: 4 x 7 mL EDTA tubes + 3 x 5 mL EDTA tubes + 2 x 4 mL no additive tubes + 1x 2,5 mL Paxgene tube (total: 53,5 mL) at a single time during the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with uncomplicated diabetes and low cardiovascular risk
  Interventions: Biological: blood sampling
- Group 2: Patients with uncomplicated diabetes and high cardiovascular risk
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — A unique venous blood sampling of 10 tubes: 4 x 7 mL EDTA tubes + 3 x 5 mL EDTA tubes + 2 x 4 mL no additive tubes + 1x 2,5 mL Paxgene tube (total: 53,5 mL) at a single time during the study

SUMMARY:
Diabetes and related complications, particularly cardiovascular disease, are associated to exacerbated inflammation, which is characterized by an activation into a pro-inflammatory status of myeloid cells including blood monocytes and tissue macrophages.

It is known that monocytes and macrophages sense, integrate and respond to their microenvironment and continually monitor the availability of nutrients in order to adapt their activity and metabolism accordingly. However, the molecular mechanisms driving their activation and switch to a pro-inflammatory phenotype in diabetes are not fully elucidated.

The Tricarboxylic Acid cycle is a nexus for multiple nutrient inputs and the generation of Tricarboxylic Acid cycle metabolites is nowadays thought to orient macrophage polarization. Reduced glutamine concentrations have been reported in patients with type 2 diabetes compared to healthy individuals. Ex vivo studies (mainly performed in rodent models) have shown that glutamine catabolism (glutaminolysis) is involved in the activation of macrophages by generating Tricarboxylic Acid cycle intermediates that promote the pro-inflammatory polarization of macrophages. Yet, the link - glutamine catabolism, monocytes polarization and diabetes-related cardiovascular complications - remains unclear.

The first phase of this project (GlutaDiab) aimed to clarify this association by quantifying glutamine metabolism in serum and monocytes activation of type 1 and type 2 diabetic patients and investigating the possible correlation with the risk of cardiovascular complications in a transversal cohort.

The GlutaDiab2 is the second phase of this project and aims to further investigate the association between glutamine metabolism and cardiovascular risk by collecting follow-up data on cardiovascular events. This longitudinal data will also address the directionality of the association between glutamine metabolism, monocytes activation and cardiovascular risk.

DETAILED DESCRIPTION:
During a scheduled hospitalization or consultation as part of the follow-up of their diabetes, additions of biological samples, which include:

A unique venous blood sampling of 10 tubes (total: 53,5 mL) at a single time during the study

ELIGIBILITY:
Inclusion Criteria:

* Person previously enroled in the GLUTADIAB study in group 1 or 2 (cf appendix 1 for GLUTADIAB inclusion criteria)

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Absence of free and informed consent
* Subject deprived of freedom, subject under a legal protective measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Type 1 and 2 diabetic patients
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
The main objective of the study is to compare the plasma concentrations of glutamine in patients at the first visit (baseline) and the risk of cardiovascular events occurring until the GlutaDiab2 visit | inclusion
  The primary endpoint is the association between plasma concentration of glutamine in each subject and cardiovascular events occurring during follow-up.

SECONDARY OUTCOMES:
To study cardiovascular events during follow-up according to glutamine metabolism in patients at baseline | inclusion
  For the analysis of study cardiovascular events during follow-up according to glutamine metabolism in patients at baseline:
  First occurrence of a cardiovascular events according to the plasma concentration of glutamate in each treatment group
To study cardiovascular events during follow-up according to glutamine metabolism in patients at baseline | inclusion
  For the analysis of study cardiovascular events during follow-up according to glutamine metabolism in patients at baseline:
  First occurrence of a cardiovascular events according to the plasma concentration of a-ketoglutarate, fumarate, and succinate in each treatment group
To study cardiovascular events during follow-up according to glutamine metabolism in patients at baseline | inclusion
  For the analysis of study cardiovascular events during follow-up according to glutamine metabolism in patients at baseline:
  First occurrence of a cardiovascular events according to the monocyte cytoplasmic concentration of a-ketoglutarate, fumarate and succinate in each treatment group
To study cardiovascular events during follow-up according to the inflammatory status in patients at baseline | inclusion
  For the analysis of the cardiovascular events during follow-up according to the inflammatory status in patients at baseline:
  First occurrence of a cardiovascular events according to the plasma concentration of VEGF (vascular endothelial growth factor) in each treatment group
To study cardiovascular events during follow-up according to the inflammatory status in patients at baseline | inclusion
  For the analysis of the cardiovascular events during follow-up according to the inflammatory status in patients at baseline:
  First occurrence of a cardiovascular events according to the plasma concentration of the proinflammatory cytokines IL-1 béta, IL-6, IL-8 and TNF-a
To study cardiovascular events during follow-up according to the inflammatory status in patients at baseline | inclusion
  For the analysis of the cardiovascular events during follow-up according to the inflammatory status in patients at baseline:
  First occurrence of a cardiovascular events according to the blood concentration of circulating PBMCs
To study cardiovascular events during follow-up according to the monocyte activation status in patients at baseline | inclusion
  First occurrence of a cardiovascular events according to the frequency of monocyte subsets
To study glutamine metabolism variations between baseline and follow-up visit according to variation in cardiovascular risk | inclusion
  To study glutamine metabolism variations between baseline and follow-up visit according to variation in cardiovascular risk In participants without cardiovascular events occurring during follow-up, cardiovascular risk will be assessed through clinical and biological data and coronary artery calcium score

CONTACTS AND LOCATIONS:
Overall Officials: Louis POTIER, Study Chair — Bichat Hospital
Locations (2):
- France (2):
  - Lariboisière hospital, Paris
  - Diabétologie, Paris

IPD SHARING:
Plan to Share IPD: No